CLINICAL TRIAL: NCT04775693
Title: Robotic Exoskeleton Gait Training During Acute Stroke Rehabilitation
Acronym: RERC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-911-16
Record Dates: First submitted 2021-02-03; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Acute
Keywords: hemiplegia; robotic; exoskeleton; gait
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Exoskeleton Device; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- RE (Experimental): Participants use the robotic exoskeleton (RE) in addition to their standard of care gait training as both an inpatient (2 days a week RE) and an outpatient (3 days a week RE).
  Interventions: Device: RE (Robotic Exoskeleton)
- SOC (Active Comparator): Participants receive standard of care gait training only as both an inpatient (at least 2 days a week) and an outpatient (at least 3 days a week).
  Interventions: Other: SOC (standard of care)
- RE/SOC (Experimental): Participants use the robotic exoskeleton (RE) in addition to their standard of care gait training as an inpatient (2 days a week RE) and standard of care only as an outpatient (at least 3 days a week).
  Interventions: Device: RE (Robotic Exoskeleton)

INTERVENTIONS:
Device: RE (Robotic Exoskeleton) — Participants will continue to receive their prescribed standard of care physical therapy/gait training. They will also utilize the robotic exoskeleton twice a week during their inpatient stay and 3 times a week for 5 weeks as an outpatient (for outpatient, only if in the RE group). The Robotic Exoskeleton is a device that will be strapped to the chest and legs and worn over the shoulders like a backpack that will assist in walking. It uses sensors and participant motion to move. A licensed physical therapist will be assisting participants as they use the device.
  Arms: RE; RE/SOC
Other: SOC (standard of care) — Traditional physical therapist driven gait training.
  Arms: SOC

SUMMARY:
The objective of this RCT is to explore the clinical, functional and neurophysiological effectiveness of RE-assisted (Robotic Exoskeleton) early intervention gait therapy in stroke patients during inpatient and outpatient stroke rehabilitation as compared to traditional gait training in three groups: 1) RE; 2) RE-Standard of Care (SOC) and 3) SOC. We will evaluate the short and long-term effects on functional mobility, clinical, neurophysiological, community participation and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors < 4 weeks from most recent stroke.
* Age: 21- 80 years
* Unilateral hemiparesis
* Medical clearance by a Kessler Institute for Rehabilitation physician.
* Be able to physically fit into the exoskeleton device.
* Be able to tolerate upright standing for 30 minutes.
* Have joint range of motion within normal functional limits for ambulation.
* Have sufficient strength to use the hemiwalker, bilateral canes or walker while wearing the RE.
* Have stable blood pressure; no diagnosis of persistent orthostatic hypotension (blood pressure drop of more than 30 millimeters of Mercury in body weight support system).
* Patient cognitive status and ability to communicate in English must be at a level consistent with that required to participate in standard motor rehabilitation, e.g. can follow directions as determined by a Kessler Institute for Rehabilitation physician or physical therapist.
* No history of injury or pathology to the unaffected limb.

Exclusion Criteria:

* Unable to physically fit within the RE: Height below 60" or above 76" and weight above 220 lbs.

  * Joint contracture or spasticity of any limb that limits normal ROM during ambulation with assistive devices.
  * Any medical issue that precludes full weight bearing and ambulation (e.g. orthopedic injuries, pain, severe spasticity).
  * Skin issues that would prevent wearing the device.
  * Pressure sore stage 2 or higher located in an area that would negatively affect weight bearing, harness fit, or therapist assistance.
  * Pre-existing condition that caused exercise intolerance.(Documented uncontrolled hypertension, coronary artery disease, cardiac arrhythmia, or congestive heart failure)
  * Hospitalization for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study.
  * Severe cognitive or psychiatric problems as well as incontinence might be contraindications to start training with a RE.
  * History of severe cardiac disease such as myocardial infarction, congestive heart failure.
  * Uncontrolled seizure disorder.
  * Uncontrolled spasticity that would interfere with walking in the RENeuromuscular or neurological pathologies (e.g., Parkinson's disease, spinal cord injury, or traumatic brain injury with evidence of motor weakness and multiple sclerosis) that will interfere with neuromuscular function, ambulation, or limit the range of motion of the lower limbs
  * Orthopedic pathologies or history that will interfere with ambulation or limit the range of motion of the lower limbs (e.g., knee replacement, fixed contractures, inflammation)
  * Pregnant as confirmed by pregnancy test.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | 6 months
  a conventional assessment measure of motor function
TUG | 6 months
  time up and go (TUG) test
BBA | 6 months
  Berg Balance Assessment (BBA)
ROM | 6 months
  range of motion (ROM)- conventional assessment performed by a physical therapist
strength | 6 months
  conventional assessment performed by a physical therapist
temporal spatial parameters | 6 months
  collected though motion capture camera system
plantar loading | 6 months
  use of shoe insoles to gather information about foot pressure
electromyography (EMG) | 6 months
  a measure of muscle activation (EMG signal) at different phases of gait cycle (swing versus double support).
SIS | 6 months
  stroke impact scale (SIS). questionnaire about quality of life post-stroke
LIFE-H | 6 months
  assessment of life habits (LIFE-H). questionnaire about quality of life post-stroke
SSQoL | 6 months
  stroke specific quality of life scale (SSQoL). questionnaire about quality of life post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Nolan, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No